CLINICAL TRIAL: NCT00253318
Title: Phase I, Open Label, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of the Combination RAD001 Plus Docetaxel in Patients With Metastatic Breast Cancer
Brief Title: RAD001 Plus Docetaxel in Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity and Lack of Efficacy
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0758; NCI-2010-00840 (Registry Identifier: NCI CTRP); NCT01825265 (obsolete NCT alias)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Neoplasm Metastasis; Breast Cancer; Docetaxel; RAD001; Taxotere
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Everolimus; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 + Docetaxel (Experimental): RAD001 30 mg orally on Days 1 and 8. Docetaxel 40 mg/m^2 intravenous (IV) over 1 hour on Day 1. Dexamethasone 8 mg orally twice daily for 3 days, starting 24 hours prior to the administration of Docetaxel.
  Interventions: Drug: Docetaxel; Drug: RAD001; Drug: Dexamethasone

INTERVENTIONS:
Drug: Docetaxel — 40 mg/m^2 IV over 1 hour on Day 1.
  Other Names: Taxotere
Drug: RAD001 — 30 mg orally on Days 1 and 8.
Drug: Dexamethasone — 8 mg orally twice daily for 3 days, starting 24 hours prior to the administration of Docetaxel.
  Other Names: Decadron

SUMMARY:
Primary:

* To assess the safety and tolerability and to find the maximum tolerated dose of the combination administration of RAD001 plus docetaxel when given to patients with metastatic breast cancer who are being considered for standard docetaxel treatment (phase I).
* To characterize the pharmacokinetics of RAD001 and docetaxel when co-administered (phase I).

Secondary:

* To determine the phosphorylation status of the components of the mTOR signaling pathway and the expression of modifiers of apoptosis in the primary breast tumors, in order to determine whether these markers can be used as predictors of sensitivity to the combination of RAD001 and docetaxel
* To determine the effect of the combination of RAD001 and docetaxel on the expression and phosphorylation of mTOR's targets in the accessible tumor tissue, in order to identify potential pharmacodynamics markers of response to this drug combination

DETAILED DESCRIPTION:
Docetaxel is a drug approved for the treatment of metastatic breast cancer in patients who are either newly diagnosed or have failed earlier chemotherapy. RAD001 is an investigational drug that has shown to have anticancer properties. It also works by weakening the immune system. RAD001 works by blocking some of the steps required for cancer growth. The researcher hopes that RAD001 may increase the anticancer activity of docetaxel.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. Blood (between 1-2 teaspoons) will be collected for routine tests. You will have scans (MRI or CT) to check on the status of your cancer as ordered by your primary physician. Women who are able to have children must have a negative blood pregnancy test. As part of the study researchers will also look at the tissue of your original cancer. Special stains will be done that will help find ways in which researchers can predict the response of your cancer to RAD001.

If you are found to be eligible to take part in this study, you will receive docetaxel by vein on Day 1 over one hour. RAD001 will be given by mouth on Days 1 and 8. RAD 001 will be given on an empty stomach or after a light meal. You will repeat this treatment every 21 days. Three (3 ) weeks equals 1 cycle.

Patients who participate on the first part of this study will be enrolled in groups of 3 at a time. The dose of RAD001 will be increased with each new group of patients. The dose of docetaxel will remain the same. The second part of the study will be using the highest dose of RAD001 and docetaxel that was found to be safe and effective during the first part of the study. (***Study did not progress to second part.***)

Dexamethasone will be given by mouth twice a day for 3 days, starting the day before you receive docetaxel. Dexamethasone helps decrease the risk of and control nausea, vomiting, and fluid retention.

Blood (between 1-2 teaspoons) will be drawn for routine tests at each visit. X-rays and scans (CT or MRI) will be done every 6 weeks to see if the tumor is responding to treatment.

After 6 cycles of the combination, docetaxel will be stopped and you will continue to take RAD001 alone. However, you may be able to take more than 6 cycles of the combination if you are not having any side effects and is found to be of benefit by your primary doctor.

Once you go off treatment, you will have a physical exam, including routine blood tests (1-2 teaspoons).

This is an investigational study. Docetaxel is approved by the FDA and commercially available for the treatment of breast cancer. RAD001 is authorized for use in research only. About 65 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of metastatic breast cancer with at least one measurable or evaluable lesion. For the phase II portion of the study patients will be required to have measurable disease. Response will be determined using the Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
3. No limit on the prior number of chemotherapies for the phase I portion of the study. No more than one prior chemotherapy regimen for the phase II portion of the study.
4. Signed informed consent to participate in the study must be obtained from patients after they have been fully informed on the nature and potential risks by the investigator with the aid of written information.
5. Adequate bone marrow function as shown by: Absolute neutrophil count (ANC) > or = 1.5 times 10(9)/L, Platelets > or = 100 times 10(9)/L, Hgb > or = 10g/dL.
6. Normal renal function as shown by serum creatinine < or = 1.5 times Upper Limit of Normal (ULN).
7. Hepatic Function Variables:

   * Bilirubin < or = ULN
   * Alkaline phosphatase < or = 5 times ULN. If alkaline phosphatase is < or = 2.5 times ULN, ALT/AST must be < or = 2.0 times ULN. If alkaline phosphatase is > 2.5 but < or = 5 times ULN, ALT/AST must be < or = 1.5 times ULN
8. Performance Status 0-2 on the World Health Organization (WHO) scale.

Exclusion Criteria:

1. Patients enrolled in the Phase I portion of the trial may have received prior docetaxel in the adjuvant or metastatic setting. Patients enrolled in the Phase II portion of the trial will not be considered eligible if they have received prior docetaxel as treatment for metastatic breast cancer. For the purposes of this protocol, patients who develop systemic metastasis < 6 months from adjuvant docetaxel will be considered to have had treatment with docetaxel for metastatic breast cancer and will be ineligible for protocol participation.
2. Patients with a history of thromboembolism within the prior 6 months or active thrombophlebitis.
3. For the phase I portion of the study, patients with grade > 2 neuropathy, for the phase II portion of the trial, patients with > or = grade 2 neuropathy.
4. For the phase I portion of the trial, patients with treated brain metastasis that are stable for 3 months will be eligible for protocol participation. However, patients with brain metastasis will be excluded from the phase II portion of the trial.
5. Patients with an uncontrolled infection.
6. Patients with a known history of HIV seropositivity.
7. Patients with an active, bleeding diathesis, or on oral anti-vitamin K medication (except patients receiving 1 mg of warfarin to prevent central venous catheter thrombosis).
8. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration).
9. Patients with impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
10. Patients who received any other investigational drugs within the preceding 30 days.
11. Patients who have received mitomycin C or nitrosourea.
12. Patients receiving anti-neoplastic therapy less than 14 days prior to entry onto this study or who have not recovered from the toxic effects of such therapy.
13. Patients who received radiation therapy within 3 weeks prior to entry on this study or who have not recovered from the toxic effects of such therapy.
14. Patients who had surgery within 2 weeks prior to entry on this study or who have not recovered from the side effects of such therapy.
15. Patients with a history of noncompliance to medical regimens.
16. Patients unwilling to or unable to comply with the protocol.
17. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A4 or patients taking lithium chloride.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of combination of RAD001 plus Docetaxel | 3 week cycles

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org